CLINICAL TRIAL: NCT01816464
Title: Immunogenicity and Safety of Trivalent Influenza Vaccine in Pregnant and Non-pregnant HIV-Uninfected Women: An Open Label Trial
Brief Title: Immunogenicity and Safety of Trivalent Influenza Vaccine in Pregnant and Nonpregnant HIV Uninfected Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Michelle Groome, Investigator, University of Witwatersrand, South Africa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MatFlu_HIVneg_preg+nonpreg
Record Dates: First submitted 2013-03-14; First posted 2013-03-22 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Influenza
Keywords: Influenza; Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trivalent Influenza Vaccine (Experimental): The formulation based on the WHO recommendation for influenza vaccines for 2013 for the Southern-hemisphere included the following vaccine strains:
  * an A/California/7/2009 (H1N1)pdm09-like virus;
  * an A/Victoria/361/2011 (H3N2)-like virus;
  * a B/Wisconsin/1/2010-like virus.
  Dose: Single Dose 0.5 mL of TIV from pre-filled syringe.
  Interventions: Biological: Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Trivalent Influenza Vaccine — The formulation based on the WHO recommendation for influenza vaccines for 2013 for the Southern-hemisphere included the following vaccine strains:
  * an A/California/7/2009 (H1N1)pdm09-like virus;
  * an A/Victoria/361/2011 (H3N2)-like virus; - a B/Wisconsin/1/2010-like virus.
  The vaccine to be used in the study in 2013 is Vaxigrip (Sanofi Pasteur), or other equivalent licensed vaccine should the latter not be available, which will be procured commercially in pre-filled syringes. Using aseptic technique, participants will be injected with 0.5 mL of TIV from pre-filled syringe.
  Other Names: Vaxigrip

SUMMARY:
The overall aim of this project is to evaluate the immunogenicity of TIV vaccination in HIV-uninfected pregnant women compared with HIV-uninfected non-pregnant women in 2013. Safety data will also be collected.THe Pregnancy outcomes and the transplacental transfer of antibodies will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: All women

(i) Documented to be HIV-1 uninfected on one assay used in the Prevention of Mother to Child Transmission (PMTCT)/ other program undertaken within 12 weeks of study enrolment.

(ii) Able to understand and comply with planned study procedures. (iii) Provides written informed consent prior to initiation of study. (iv) Women age ≥ 18 years to < 39 years.

Inclusion Criteria: pregnant women

(i) Gestational age ≥20 weeks to <36 weeks documented by the approximate date of the last menstrual period and corroborated by physical exam and sonar report if available.

Exclusion Criteria:

Exclusion Criteria: All women

(i) Receipt of TIV, other than through the study, during the current influenza season documented by medical history or record.

(ii) Receipt of any live licensed vaccine ≤ 28 days or any other vaccine (except for tetanus toxoid vaccine) ≤ 14 days prior to study-vaccine.

(iii) Receipt of a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) ≤ 28 days prior to vaccination in this study, or expects to receive another non-licensed agent before delivery unless study approval is obtained.

(iv) Any significant (in the opinion of the site investigator) acute illness and/or oral temperature greater than or equal to 38 degrees C ≤ 24 hours prior to study entry.

(v) Use of anti-cancer systemic chemotherapy or radiation therapy ≤ 48 weeks of study enrollment, or has immunosuppression as a result of an underlying illness or treatment.

(vi) Long term use of glucocorticoids, including oral or parenteral prednisone ≥ 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) ≤ 12 weeks of study entry, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) ≤ 12 weeks before study entry (nasal and topical steroids are allowed).

(vii) Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) ≤ 12 weeks prior to enrollment in this study or is scheduled to receive immunoglobulin or other blood products (with the exception of Rho D immune globulin) during pregnancy or for the first 24 weeks after delivery.

(viii) Receipt of immune mediators ≤ 12 weeks before enrollment. (ix) Uncontrolled major psychiatric disorder. (x) History of a severe adverse reaction to previous TIV. (xi) Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Exclusion Criteria: pregnant women

(i) Receipt of corticosteroids for preterm labor ≤ 14 days before study entry. (ii) Pregnancy complications (in the current pregnancy) such as pre-term labor, hypertension (Blood Pressure (BP) >140/90 in the presence of proteinuria or BP >150/100, with or without proteinuria or currently on antihypertensive medication) or pre-eclampsia.

-

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Compare the immunogenicity of Trivalent Influenza Vaccine (TIV) in pregnant compared to non-pregnant Human Immunodeficiency Virus (HIV)-uninfected women. | one month post-vaccination
  Hemagglutination inhibition assays (HAI)will be performed to assess the immunogenicity of TIV. In this study we will use the following definitions to assess the humoral immune response to TIV: HAI titers <1:10 = seronegative; HAI titers ≥1:10 = seropositive; HAI titers ≥1:40 = sero-protective titers; and sero-conversion will be defined as HAI titers from <1:10 to ≥1:40 or ≥4-fold increase if pre-vaccination titers were ≥1:10.
Evaluate the immunogenicity of Trivalent Influenza Vaccine (TIV) in pregnant Human Immunodeficiency Virus (HIV)-uninfected women at time of delivery | one week post delivery for the pregnant cohort
  Hemagglutination inhibition assays (HAI)will be performed to assess the immunogenicity of TIV. In this study we will use the following definitions to assess the humoral immune response to TIV: HAI titers <1:10 = seronegative; HAI titers ≥1:10 = seropositive; HAI titers ≥1:40 = sero-protective titers; and sero-conversion will be defined as HAI titers from <1:10 to ≥1:40 or ≥4-fold increase if pre-vaccination titers were ≥1:10.

SECONDARY OUTCOMES:
Determine the impact of vaccination on T-cell activation and regulatory B and T cells subpopulations in pregnant and non-pregnant women. | one month post vaccination and one week post delivery in pregnant cohort
  T-lymphocyte activation assays will be performed using state-of-the art polychromatic flow cytometry. The T- and B-cell phenotypes are assessed by flow cytometry using freshly thawed Peripheral Blood Mononuclear Cells (PBMC). Cells are stained using monoclonal antibodies against the comparator molecules
2.2.2. Determine the impact of vaccination on cell-mediated immune responses to each influenza strain in HIV-uninfected pregnant and non-pregnant women | one month post vaccination
  Interferon (IFN)- Enzyme Linked Immuno Spot (ELISPOT) responses will be assessed on fresh PBMCs. PBMCs will be separated and stimulated with influenza virus corresponding to the vaccine strains.Spots will be visualized with a ELISPOT plate reader. Results will be reported as Spot Forming Cells (SFC) /106 PBMCs.
Determine the dynamics of transplacental transfer of maternal Hemagglutinin (HA) antibodies to their newborns. | one week post delivery in pregnant cohort
  The study will assess the effect of TIV administration during pregnancy on transplacental influenza-specific antibody transfer to the fetus. HAI titers will be measured in infants within one week of birth. Using the 1:40 HAI titer as a defining threshold of protection against wild type influenza, we will determine the proportion of infants protected against influenza at birth.
Determine antibodies against TIV present in breast milk | in week post delivery
  Influenza specific antibodies measures by HAI titres in the breastmilk will be measured. Mothers will express breastmilk into sterile containers to collect the samples.
Compare local and systemic solicited reactions to TIV in pregnant and non-pregnant HIV-uninfected women. | one month post vaccination
  Participants will remain in the clinic for at least 30 minutes after vaccination so that clinic personnel can observe for any potential adverse reactions to the vaccine.
  Report of vaccine-related local (redness, swelling, tenderness, itching,) and systemic (fever, malaise, myalgia, nausea, headache, rash) adverse events will be solicited at day 7 and day 28 by means of a participant diary card. Serious Adverse Events (SAEs) will be reported.
Describe safety outcome measures (maternal and foetal) of TIV-vaccination of HIV-uninfected pregnant women. | one month post vaccination and one week post delivery in pregnant cohort
  Safety and tolerability of the study vaccine will be monitored by means of Adverse Events (AEs) and toxicity reports presenting laboratory and clinical data. The data to be reviewed by the protocol team will be pooled across treatment arms.In addition to monthly toxicity reviews by the Core Team, the study will be monitored by a Safety Monitoring Committee (SMC). The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events is used
Describe obstetric outcomes in HIV-uninfected pregnant women who received TIV | one week post delivery in pregnant cohort
  Data will be collected from birth records including low birth weight (<2 500 g), premature delivery (<37 weeks), emergency caesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, PHD, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Nrf/Dst Vpd Rmpru, Soweto, GP, South Africa